CLINICAL TRIAL: NCT03180671
Title: The Effectiveness of Anterior Deprogrammers as a Tool for Reducing Pain and Masticatory Muscles Tension
Brief Title: Anterior Deprogrammers for Reducing Pain and Masticatory Muscles Tension
Acronym: Deprogrammer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lukasz Adamczyk (Other)
Responsible Party: Sponsor-Investigator, Lukasz Adamczyk, Principal investigator, Wroclaw Medical University
Organization: Wroclaw Medical University (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: Anterior Deprogrammers
Record Dates: First submitted 2017-06-03; First posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Temporomandibular Disorders
Keywords: anterior deprogrammer; muscle pain; centric relation
MeSH Terms: conditions — Temporomandibular Joint Disorders; Myalgia | interventions — Occlusal Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Group 1 Control (No Intervention): Counselling with explanation of preventive procedures.
- Group 2 deprogramer Sliding Guide (Active Comparator): Intervention using the Deprogrammer Sliding Guide for 12-15 minutes.
  Interventions: Device: Deprogramer Sliding Guide
- Group 3 deprogrammer Dawson B-Splint (Active Comparator): Intervention using the Dawson B-Splint for 7 days with breaks for eating/drinking and oral hygiene procedures.
  Interventions: Device: Deprogrammer Dawson B-Splint
- Group 4 deprogrammer Kois (Active Comparator): Intervention using the Kois deprogrammer for 14 days with breaks for eating/drinking and oral hygiene procedures.
  Interventions: Device: Deprogrammer Kois

INTERVENTIONS:
Device: Deprogramer Sliding Guide — Use of the intraoral device.
  Other Names: Occlusal splint
  Arms: Group 2 deprogramer Sliding Guide
Device: Deprogrammer Dawson B-Splint — Use of the intraoral device.
  Other Names: Occlusal splint
  Arms: Group 3 deprogrammer Dawson B-Splint
Device: Deprogrammer Kois — Use of the intraoral device.
  Other Names: Occlusal splint
  Arms: Group 4 deprogrammer Kois

SUMMARY:
The study will be conducted in four groups of 20 patients in age of 20-30 years with complete dentition or single tooth loss in lateral regions, with masticatory muscle pain in the history or during examination and overuse and/or chronic tensing of the masticatory muscles. Patients will be randomly assigned to the groups.

Each person will be measured twice before and after use of selected anterior deprogrammer. The following assessment tools will be applied:

* surface electromyography of masseter and temporal muscles,
* intraoral pin-supported registration to draw a gothic arch.

Measurements will be made before and after intervention to assess the effect of anterior deprogrammer application on the tone of the selected masticatory muscles and condyles position in mandibular fossa. The first group (control) will be counsel with an explanation of the pathomechanism of masticatory muscles pain and preventive principles. In the second group, the Sliding Guide will be used for a period of 12-15 minutes, in the third Dawson B-Splint for 7 days, and in the fourth Kois deprogrammer for 14 days. Devices in group 3 and 4 will be used by patients for 24 hours a day, with breaks for oral hygiene procedures and eating/drinking.

The aim of the study is to evaluate the effectiveness of selected anterior deprogrammers.

ELIGIBILITY:
Inclusion Criteria:

* age 20-30 years old
* complete dentition or single tooth loss in the lateral regions
* no severe systemic diseases
* masticatory muscle pain in the history or during examination
* increased masticatory muscles tension

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Electromyography | 2 min
  Examination of masseters and temporal muscles tension

SECONDARY OUTCOMES:
Centric relation | 5 min
  Registration of centric relation with Sm-Registration-set (intraoral pin-supported registration)

CONTACTS AND LOCATIONS:
Overall Officials: Mieszko Wieckiewicz, DMD, MSc, PhD, Study Chair — Wroclaw Medical University; Lukasz Adamczyk, DMD, Principal Investigator — Dental Practice
Locations (1):
- Dental Practice, Tarnów, Poland

IPD SHARING:
Plan to Share IPD: No